CLINICAL TRIAL: NCT02055911
Title: Retinal Ganglion Cell Function After Repeated Intravitreous Ranibizumab in Diabetic Macular Edema
Brief Title: Retinal Ganglion Cell Function After Intravitreous Ranibizumab in Patients With Diabetic Macular Edema
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Mauricio Maia, Professor, Federal University of São Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Retinal Ganglion Cell_DME
Record Dates: First submitted 2014-02-03; First posted 2014-02-05 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2014-02

CONDITIONS: Diabetic Macular Edema
Keywords: diabetic macular edema; intravitreal ranibizumab; f retinal ganglion cell
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ranibizumab (Experimental): monthly ranibizumab (0,5 mg injected intravitreally in a standard fashion) until maximum visual acuity (VA) is achieved and remains stable for three consecutive months (for a minimum of 3 initial injections).
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — monthly ranibizumab (0,5 mg injected intravitreally in a standard fashion) until maximum visual acuity (VA) is achieved and remains stable for three consecutive months (for a minimum of 3 initial injections).
  Other Names: Lucentis

SUMMARY:
To evaluate the safety of intravitreal ranibizumab repeated injections in patients with diabetic macular edema regarding maintenance of retinal ganglion cell function.

DETAILED DESCRIPTION:
* Ranibizumab can be a safe treatment for diabetic macular edema regarding maintenance of retinal ganglion cell function after repeated intravitreal injections.
* To evaluate the safety of intravitreal ranibizumab repeated injections in patients with diabetic macular edema regarding maintenance of retinal ganglion cell function.
* The primary endpoint for the study will be the changes in full-field and focal macular photopic negative response (PhRN) amplitude (in µV) over time, from baseline to month 12.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, older than 18 years, who have signed an informed consent.
* Patients with Type 1 or Type 2 diabetes mellitus and prior diagnosis of diabetic macular edema (DME), who had not undergone any previous treatment, either pharmacological or laser photocoagulation.
* Patients with visual impairment due to DME whom, in the opinion of the investigator, would benefit from treating with IVR.

Exclusion Criteria:

* Known hypersensitivity to ranibizumab or any of its components.
* Previous participation in any clinical studies of investigational drugs within 1 month
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, including women whose career, lifestyle, or sexual orientation precludes intercourse with a male partner and women whose partners have been sterilized by vasectomy or other means, UNLESS they are using two birth control methods. The two methods can be a double barrier method or a barrier method plus a hormonal method. Adequate barrier methods of contraception include: diaphragm, condom (by the partner), intrauterine device (copper or hormonal), sponge or spermicide. Hormonal contraceptives include any marketed contraceptive agent that includes an estrogen and/or a progestational agent.
* Pregnant or nursing (lactating) women.
* Inability to comply with study or follow-up procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2015-03 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
focal macular changes in full-field and photopic negative response (PhRN) amplitude (in µV) | at Baseline and Months 3, 6, 9, 12
  The photopic negative response (PhNR) of the full-field cone electroretinograms (ERGs) is a functional indicator of retinal ganglion. The PhNR consists of a negative-going wave that follows the photopic cone b wave. The PhNR is selectively attenuated in patients with optic nerve disease and glaucoma, indicating that the PhNR can be an objective functional measure reflecting the sum of the total response of the retinal ganglion cells in the entire retina.

SECONDARY OUTCOMES:
The mean change in BCVA | monthly, from baseline to Month 12
  The mean change in best corrected visual acuity (BCVA) from baseline to month 12
the mean change in central macular thickness (CMT) | monthly, from baseline to Month 12
  To assess the mean change in central macular thickness (CMT), measured in spectral-domain optical coherence tomography (SD-OCT) from baseline to month 12

OTHER OUTCOMES:
assess adverse events | monthly, from Month 1 to Month 12
  To assess adverse events during the twelve months of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Mauricio Maia, MD, Principal Investigator — UNIFESP / HOSPITAL SÃO PAULO
Locations (1):
- Dept of Ophthalmology - UNIFESP/Hospital São Paulo, São Paulo, São Paulo, Brazil